CLINICAL TRIAL: NCT02205710
Title: Adaptive Cognitive Training in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: M16-14-018
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2017-08

CONDITIONS: Mild Cognitive Impairment; Mild to Moderate Dementia; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Computerized cognitive training (Experimental): Series of gamified tasks.
  Interventions: Other: Computerized cognitive training
- Computerized game training (Placebo Comparator): Series of gamified tasks.
  Interventions: Other: Computerized games

INTERVENTIONS:
Other: Computerized cognitive training
  Other Names: Activate
  Arms: Computerized cognitive training
Other: Computerized games
  Arms: Computerized game training

SUMMARY:
Cognitive training has emerged as a promising method to maintain, enhance, and rehabilitate cognitive function in older adults and individuals with dementia. In recent years, such training has become particularly appealing in the clinical context, with many paradigms aimed specifically at adults experiencing various stages of cognitive decline due to Mild Cognitive Impairment, Alzheimer's disease, and vascular dementias. However, basic questions remain. For example, uncertainty persists regarding factors that influence observed improvements as well as the conditions that would maximize transfer and sustainability of training effects. The objective of this study is to evaluate factors that may maximize the benefits of computerized cognitive training in older adults.

DETAILED DESCRIPTION:
The study involves 25 sessions of an adaptive cognitive training program, completed over 5 weeks. Pre and post training assessments will evaluate any near and far transfer effects of training.

ELIGIBILITY:
Inclusion Criteria:

* English as the maternal or primary spoken language.
* Good self-reported health (i.e., no cerebro-, or cardio-vascular disease or neurological disease).
* Normal or corrected-to-normal vision and hearing.

Exclusion Criteria:

* Poor hearing or vision
* Inadequate understanding of the English language

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in ratings on cognitive training survey | Baseline, week 5
  This survey aims to assess participant perceptions on cognitive training, and includes a series of related questions, rated on a scale of 1-7.
Change in neural activity | Baseline, week 5
  We will measure resting state as well as task-related EEG responses to determine the effects of cognitive training at the neural level.
Change in performance on neuropsychological tests | Baseline, week 5
  Using a set of standard neuropsychological evaluations, we will measure changes in attention, memory, and executive function following cognitive training.

SECONDARY OUTCOMES:
Change in ratings of psychological wellbeing | Baseline, week 5
  We will use standardized questionnaires to assess quality of life, in order to measure the influence of cognitive training on factors related to wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Davidson, PhD, Principal Investigator — University of Ottawa; Sheida Rabipour, MSc, Study Director — University of Ottawa
Locations (1):
- Bruyere Continuing Care, Ottawa, Ontario, Canada